CLINICAL TRIAL: NCT06181981
Title: Longitudinal Evaluation of Leucoaraiosis Using Multimodal MRI With Fingerprinting Technique
Brief Title: Leucoaraiosis and Multimodal MRI With Fingerprinting Technique
Acronym: LEUKOPRINT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Lille Catholic University (Other)
Collaborators: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: RNIPH-2022-03
Record Dates: First submitted 2023-12-13; First posted 2023-12-26 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Leukoaraiosis; Magnetic Resonance Imaging
Keywords: Leukoaraiosis; Magnetic Resonance Imaging; White Matter Hyperintensities (WMH); Normal Appearing White Matter (NAWM)
MeSH Terms: conditions — Leukoaraiosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- incidental Leukoaraiosis (LA): Eligible patients in the incidental LA group will be pre-identified by the radiologist at the time of the 3T MRI or CT scan, and recruited by the neurologist at their first routine neurology consultation in the days following the MRI.
  Interventions: Diagnostic Test: MRI fingerprinting
- LA and ischemic stroke: Eligible patients in the LA + ischemic stroke group will be recruited by the neurologist during hospitalization for ischemic stroke
  Interventions: Diagnostic Test: MRI fingerprinting
- LA and intracerebral hemorrhage: Eligible patients in the LA + intracerebral hemorrhage group will be recruited by the neurologist during hospitalization
  Interventions: Diagnostic Test: MRI fingerprinting

INTERVENTIONS:
Diagnostic Test: MRI fingerprinting — This method allows to get quantitative magnetic resonance imaging for the simultaneous measurement of multiple tissue properties in a single, time-efficient acquisition

SUMMARY:
Leukoaraiosis (LA) corresponds to an alteration of the encephalic white matter, linked to chronic hypoxia. Its pathophysiology, which has been partially elucidated, is underpinned by chronic changes in the walls of small-caliber perforating arteries, leading to chronic hypoperfusion of the white matter, associated with dysfunction of the blood-brain barrier. In affected areas, this process leads to myelin rarefaction, axonal loss, perivascular alterations and the appearance of cavitation zones. Its existence is mainly linked to the presence of vascular risk factors, most notably arterial hypertension.

MR fingerprinting is an innovative Magnetic resonance Imaging (MRI) technique allowing to obtain a multiparametric MRI sequence in a non-invasively way and in a single acquisition, generating not only multiple contrasts, but also absolute longitudinal relaxation time (T1) and transverse relaxation time (T2) mappings (T1 and T2 mapping). However, the prognostic role of these T2 values, in terms of ischemic, hemorrhagic and cognitive risk, has never been studied. The objective of this study is to study and compare changes in T1 and T2 values of White Matter Hyperintensities (WMH) and Normal Appearing White Matter (NAWM) in subjects with LA.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 40 years of age
* Suffering from leucoaraiosis
* Diagnosed via cerebral MRI or CT scan performed by the St Philibert Hospital imaging department

For the groups:

* incidental LA (patients included in group 1): on the MRI, FLAIR images showed the presence of hyperintense white matter lesions, assessed at a minimum FAZEKAS grade 2+2, the origin of which was related to small artery disease discovered incidentally or during acute management in GHICL's neurovascular intensive care unit. The CT scan revealed hypodense patches of deep periventricular white matter, also of minimal Fazekas grade 2+2.
* LA and ischemia (patients included in group 2): on the MRI, FLAIR images show the presence of hyperintense white matter lesions with an extent assessed at a minimum grade of FAZEKAS 2+2: their origin is related to small artery disease discovered during acute management of cerebral ischemia in the GHICL's Neurovascular Intensive Care Unit.
* LA and cerebral hemorrhage (patients included in group 3): on the MRI, FLAIR images show the presence of hyperintense white matter lesions of minimal FAZEKAS grade 2+2: their origin is related to small artery disease discovered during the acute management of a cerebral hemorrhage, in the GHICL's Neurovascular Intensive Care Unit.

Exclusion Criteria:

* Claustrophobia preventing MRI scan
* MRI contraindication
* White matter lesions with diagnosis not formally established, doubtful, multifactorial or related to a differential diagnosis
* Patients with dementia or pathology that precludes longitudinal follow-up
* Institutionalized patients
* Agitation not allowing MRI to be performed
* Pregnant women
* Patients under guardianship
* Patients objecting the use of their data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient over 40 years of age suffering from leucoaraiosis diagnosed via cerebral MRI or CT scan performed by the St Philibert Hospital (GHICL) imaging department
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2022-11-14 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
T1 (seconds) | 30 months
  T1 will be measured by three-dimensional, magnetization-prepared rapid gradient-echo (3D MP-RAGE) imaging
T2 (milliseconds) | 30 months
  T2 will be measured by three-dimensional segmented echo-planar-imaging (3D T2 EPI)

SECONDARY OUTCOMES:
Correlation coefficient and its 95% confidence interval between WMH T1 and T2 values, and WHM lesion volume. | 30 months
  Correlation between T1 and T2 values and WHM lesion volume will be assessed by Pearson's or Spearman's correlation coefficient in the absence of normality, and its 95% confidence interval. Correlation will be considered very good if |ρ| > 0.8; good if |ρ| is between 0.61 and 0.8; moderate if |ρ| is between 0.6 and 0.41; poor otherwise.
Correlation coefficient and its 95% confidence interval between T1 and T2 values of WMH and NAWM, lesion volume of WMH, and number of microbleeds | 30 months
  Correlation between T1 and T2 values and WHM lesion volume will be assessed by Pearson's or Spearman's correlation coefficient in the absence of normality, and its 95% confidence interval. Correlation will be considered very good if |ρ| > 0.8; good if |ρ| is between 0.61 and 0.8; moderate if |ρ| is between 0.6 and 0.41; poor otherwise.

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien VERCLYTTE, MD, Study Director — Groupement des Hopitaux de l'institut catholique de Lille
Locations (1):
- Grupement des Hôpitaux de l'Institut Catholique de Lille, Lomme, France

IPD SHARING:
Plan to Share IPD: No